CLINICAL TRIAL: NCT01894022
Title: An Open-label Extension Study of the Long-term Safety, Tolerability and Efficacy of Ambrisentan in Subjects With Inoperable Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Brief Title: A Open Label Study to Assess the Long-term Safety, Tolerability and Efficacy of Ambrisentan in Subjects With Inoperable Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Acronym: AMBER II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116457
Record Dates: First submitted 2013-07-03; First posted 2013-07-09 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Hypertension
Keywords: Inoperable chronic thromboembolic pulmonary hypertension, endothelin receptor antagonist
MeSH Terms: conditions — Hypertension | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ambrisentan Arm (Experimental): All subjects will receive ambrisentan initially at a dose of 5 mg once daily (OD). Based on the investigator's best judgment, the subject may continue on 5 mg OD, or be up-titrated to 10 mg OD. The dose may also be adjusted back to 5 mg OD at investigator discretion.
  Interventions: Drug: Ambrisentan 5 mg

INTERVENTIONS:
Drug: Ambrisentan 5 mg — Round, white, film-coated, immediate-release tablets, containing 5 mg ambrisentan. Subjects will be dosed orally once daily. Subjects may receive 5mg, or 10 mg of ambrisentan OD.

SUMMARY:
This is an open label, long term extension to Study AMB115811. All subjects may remain in the extension study for a minimum of 18 months. Beyond the 18-month period, subjects may continue in the extension study until one of the following: the product is approved locally for use in inoperable CTEPH patients; development for use in the CTEPH population is discontinued or product is not approved by the local regulatory authorities; or the investigator decides to discontinue the subject or subject decides to discontinue from the study. The primary purpose of this study is to provide clinically relevant information on the long term safety of ambrisentan in subjects with inoperable CTEPH.

ELIGIBILITY:
Inclusion Criteria:

* Have been randomized to the protocol for AMB115811 and have met one of the following: Completed the Week 16 visit in AMB115811; Or Prematurely withdrew from AMB115811 for whatever reason (where investigational product [IP] has been stopped due to safety or efficacy reasons, the subject may still enter into the open label study regardless of what treatment they are receiving [other treatments will not be supplied by the sponsor]. The investigator will decide whether or not the subject will receive the IP
* Subject is able and willing to give written informed consent. As part of the consent, female subjects of childbearing potential will be informed of the risk of teratogenicity and will need to be counseled in a developmentally appropriate manner on the importance of pregnancy prevention; and male subjects will need to be informed of potential risk of testicular tubular atrophy and aspermia.
* Specific information regarding warnings, precautions, contraindications, adverse events, and other pertinent information on the GSK investigational product or other study treatment that may impact subject eligibility is provided in the Investigators Brochure and product label for PAH indication.
* In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Subject meeting any of the following criteria must not receive ambrisentan, however may still be followed-up as part of the study and be treated according to best clinical practice as decided by the investigator:
* Subject has a known hypersensitivity to the Investigational Products, the metabolites, or formulation excipients
* Female subjects who are pregnant or breastfeeding or no-longer agree to comply with using effective contraception as defined in the protocol.
* Subjects with alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >= 3x Upper limit of normal (ULN)
* Subjects with bilirubin >= 2xULN (>35% direct bilirubin)
* Subjects with severe renal impairment (estimated creatinine clearance <30 millilitre per minute (mL/min) assessed within the previous 45 days) at the point of transition from Study AMB115811
* Subject has moderate - severe hepatic impairment (Child-Pugh class B-C with or without cirrhosis) at the point of transition from study AMB115811
* Subject with clinically significant fluid retention in the opinion of the investigator
* Subject with clinically significant anemia in the opinion of the investigator
* Subjects who are to enter another clinical trial or be treated with another investigational product after exiting Study AMB115811.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2015-11-18 (Actual); Study Completion 2015-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (45):
- United States (2):
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Dallas, Texas
- Argentina (4):
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Corrientes
  - GSK Investigational Site, Santa Fe
- Austria (3):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Vienna
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, London, Ontario
- China (4):
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
- GSK Investigational Site, Prague, Czechia
- Germany (7):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
- Israel (2):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Zrifin
- Japan (7):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Monterrey NL, Nuevo León, Mexico
- GSK Investigational Site, Amsterdam, Netherlands
- Russia (2):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Tomsk
- GSK Investigational Site, Riyadh, Saudi Arabia
- GSK Investigational Site, Seoul, South Korea
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Seville
- United Kingdom (3):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Clydebank
  - GSK Investigational Site, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, long-term extension study to the double-blind, placebo-controlled study AMB115811 (NCT01884675). Only those participants (par.) in study AMB115811 were eligible for enrollment in this study. The planned duration was a minimum of 18 months, but the study was terminated due to futility of enrollment in study AMB115811.
Pre-assignment Details: Out of the 33 participants randomized (16 participants in the Placebo arm and 17 in the Ambrisentan arm) in study AMB115811, a total of 19 participants were enrolled in this extension study.
Groups:
- Previous Placebo: Participants received placebo tablet once daily (OD) for 16 weeks in study AMB115811. Upon enrollment in the extension study AMB116457, participants received ambrisentan 5 milligrams (mg) tablet OD. The dose could be up-titrated to ambrisentan 10 mg OD or adjusted back to ambrisentan 5 mg OD.
- Previous Ambrisentan: Participants received ambrisentan 5 mg tablet OD for 16 weeks in study AMB115811. Upon enrollment in the extension study AMB116457, participants continued to receive ambrisentan 5 mg OD. The dose could be up-titrated to ambrisentan 10 mg OD or adjusted back to ambrisentan 5 mg OD.
Period: Overall Study
Arm/Group | Previous Placebo | Previous Ambrisentan
Started | 9 | 10
Completed | 0 | 0
Not Completed | 9 | 10
Not completed — Death | 1 | 0
Not completed — Adverse Event, non-fatal | 1 | 0
Not completed — Study Closed/terminated | 7 | 10

BASELINE CHARACTERISTICS:
Population: Participant characteristics at the start of the extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Previous Placebo | Previous Ambrisentan | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 63.0 (7.99) [58.0 to 69.0] | 61.0 (11.71) [47.0 to 66.0] | 63.0 (10.06) [54.0 to 69.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 3 | 6 | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 2 | 1 | 3
  Asian - Japanese Heritage | 2 | 1 | 3
  White - White/Caucasian/European Heritage | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect. Refer to the general AE/SAE module for a list of AEs and SAEs. Participant's final visit in Study AMB115811 was used as the entry visit of this open-label extension study. Safety (Extension) Population: all participants who enrolled and took at least one dose of study treatment during the extension study.
Time Frame: From entry visit of the extension study up to approximately 16 months
Population: Safety (Extension) Population
Measure: Number; unit: Participants
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 10
Participants
  Any AE | 8 | 6
  Any SAE | 3 | 0

2. Primary Outcome: Change From Study AMB115811 Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils (Absolute Neutrophil Count [ANC]), Platelet Count, and White Blood Cell (WBC) Count at the Indicated Time Points
Description: Hematology parameters were assessed at Entry visit of the extension study, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, and end of study. Change from study AMB115811 Baseline in basophils, eosinophils, lymphocytes, monocytes, total neutrophils (ANC), platelet count, and WBC count are summarized. AMB115811 Baseline is the last value recorded on or prior to start of study treatment in that study. Change from AMB115811 Baseline was calculated as the value at the indicated visit minus the Baseline value. Participant's final visit in Study AMB115811 was used as the entry visit of this open-label extension study. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). NA indicates that data were not available.
Time Frame: Baseline from study AMB115811; Entry visit of the extension study; Months 1, 3, 6, 9, 12, 15; and End of Study (assessed up to approximately 16 months)
Population: Safety (Extension) Population
Measure: Median (Inter-Quartile Range); unit: Giga per Liter (GI/L)
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 10
Giga per Liter (GI/L)
  Basophils, Entry visit, n=9, 10 | -0.010 [-0.020 to 0.000] | 0.000 [-0.010 to 0.010]
  Basophils, Month 1, n=7, 10 | -0.010 [-0.010 to 0.000] | 0.000 [-0.020 to 0.000]
  Basophils, Month 3, n=7, 8 | -0.010 [-0.020 to 0.010] | 0.000 [-0.010 to 0.020]
  Basophils, Month 6, n=5, 6 | 0.000 [-0.020 to 0.000] | 0.000 [-0.010 to 0.030]
  Basophils, Month 9, n=2, 5 | -0.025 [-0.040 to -0.010] | -0.010 [-0.020 to -0.010]
  Basophils, Month 12, n=1, 3 | -0.020 [-0.020 to -0.020] | 0.000 [-0.020 to 0.010]
  Basophils, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -0.010 [-0.010 to -0.010]
  Basophils, End of study, n=8, 9 | -0.005 [-0.025 to 0.015] | 0.000 [0.000 to 0.000]
  Eosinophils, Entry visit , n=9,10 | -0.010 [-0.090 to 0.040] | 0.005 [-0.090 to 0.030]
  Eosinophils, Month 1, n=7, 10 | -0.020 [-0.030 to 0.010] | -0.025 [-0.060 to 0.030]
  Eosinophils, Month 3, n=7, 8 | -0.030 [-0.050 to 0.020] | -0.005 [-0.055 to 0.075]
  Eosinophils, Month 6, n=5, 6 | 0.020 [-0.030 to 0.110] | -0.035 [-0.070 to 0.000]
  Eosinophils, Month 9, n=2, 5 | 0.155 [-0.040 to 0.350] | -0.020 [-0.020 to 0.150]
  Eosinophils, Month 12, n=1, 3 | -0.120 [-0.120 to -0.120] | 0.150 [-0.060 to 0.270]
  Eosinophils, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 0.190 [0.190 to 0.190]
  Eosinophils, End of study, n=8,9 | -0.020 [-0.055 to 0.035] | 0.010 [-0.030 to 0.030]
  Lymphocytes, Entry visit , n=9,10 | -0.050 [-0.160 to 0.190] | -0.090 [-0.470 to 0.000]
  Lymphocytes, Month 1, n=7, 10 | -0.190 [-0.460 to 0.140] | -0.225 [-0.270 to 0.080]
  Lymphocytes, Month 3, n=7, 8 | -0.040 [-0.180 to 0.240] | -0.215 [-0.795 to 0.185]
  Lymphocytes, Month 6, n=5, 6 | -0.250 [-0.340 to -0.170] | -0.110 [-1.030 to -0.010]
  Lymphocytes, Month 9, n=2, 5 | -0.075 [-0.380 to 0.230] | -0.360 [-0.490 to -0.090]
  Lymphocytes, Month 12, n=1, 3 | -0.090 [-0.090 to -0.090] | -0.260 [-0.280 to 0.480]
  Lymphocytes, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -0.730 [-0.730 to -0.730]
  Lymphocytes, End of study, n=8,9 | -0.090 [-0.280 to 0.005] | -0.230 [-0.390 to 0.080]
  Monocytes, Entry visit, n=9, 10 | -0.060 [-0.090 to 0.050] | -0.055 [-0.150 to 0.010]
  Monocytes, Month 1, n=7, 10 | 0.000 [-0.050 to 0.060] | 0.000 [-0.170 to 0.130]
  Monocytes, Month 3, n=7, 8 | 0.010 [-0.080 to 0.220] | -0.035 [-0.175 to 0.025]
  Monocytes, Month 6, n=5, 6 | 0.080 [0.030 to 0.100] | -0.035 [-0.200 to 0.050]
  Monocytes, Month 9, n=2, 5 | 0.075 [-0.130 to 0.280] | 0.060 [-0.100 to 0.200]
  Monocytes, Month 12, n=1, 3 | 0.010 [0.010 to 0.010] | -0.100 [-0.140 to 0.060]
  Monocytes, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 0.130 [0.130 to 0.130]
  Monocytes, End of study, n=8, 9 | -0.005 [-0.110 to 0.105] | 0.030 [-0.090 to 0.100]
  Total Neutrophils, Entry visit, n=9, 10 | -0.390 [-0.550 to 0.840] | -0.595 [-1.060 to 0.830]
  Total Neutrophils, Month 1, n=7,10 | 0.220 [-1.450 to 0.530] | -0.550 [-1.000 to 0.320]
  Total Neutrophils, Month 3, n=7, 8 | 0.190 [-0.120 to 0.450] | -0.675 [-0.965 to -0.085]
  Total Neutrophils, Month 6, n=5, 6 | 0.150 [0.040 to 0.290] | -0.285 [-0.450 to -0.250]
  Total Neutrophils, Month 9, n=2, 5 | -1.135 [-1.720 to -0.550] | -0.590 [-0.810 to 0.610]
  Total Neutrophils, Month 12, n=1, 3 | 1.730 [1.730 to 1.730] | -0.290 [-0.780 to -0.230]
  Total Neutrophils, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -0.940 [-0.940 to -0.940]
  Total Neutrophils, End of study, n=8, 9 | -0.025 [-0.435 to 0.520] | -0.740 [-1.390 to -0.250]
  Platelet count, Entry visit , n=9, 9 | -7.0 [-10.0 to 5.0] | -7.0 [-40.0 to 19.0]
  Platelet count, Month 1, n=7, 10 | -16.0 [-31.0 to 5.0] | -1.5 [-29.0 to 26.0]
  Platelet count, Month 3, n=7, 8 | -9.0 [-34.0 to 7.0] | 17.0 [-8.0 to 28.0]
  Platelet count, Month 6, n=5, 6 | -17.0 [-18.0 to -8.0] | -2.0 [-27.0 to 7.0]
  Platelet count, Month 9, n=2, 5 | -11.0 [-20.0 to -2.0] | -6.0 [-21.0 to 8.0]
  Platelet count, Month 12, n=1, 3 | -78.0 [-78.0 to -78.0] | -9.0 [-34.0 to 11.0]
  Platelet count, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -49.0 [-49.0 to -49.0]
  Platelet count, End of study, n=8, 9 | -5.0 [-53.0 to 9.5] | 12.0 [-4.0 to 14.0]
  WBC count, Entry visit, n=9, 10 | -0.20 [-1.40 to 0.90] | -0.65 [-1.60 to 0.60]
  WBC count, Month 1, n=7, 10 | -0.10 [-1.50 to 0.50] | -0.50 [-1.10 to -0.20]
  WBC count, Month 3, n=7, 8 | 0.20 [-0.40 to 0.80] | -1.10 [-1.65 to -0.15]
  WBC count, Month 6, n=5, 6 | 0.10 [0.00 to 0.20] | -0.55 [-1.50 to -0.30]
  WBC count, Month 9, n=2, 5 | -1.00 [-1.10 to -0.90] | -0.60 [-1.10 to 0.30]
  WBC count, Month 12, n=1, 3 | 1.50 [1.50 to 1.50] | -0.70 [-0.80 to 0.30]
  WBC count, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -1.40 [-1.40 to -1.40]
  WBC count, End of study, n=8, 9 | -0.25 [-0.60 to 0.60] | -1.00 [-1.40 to -0.50]

3. Primary Outcome: Change From Study AMB115811 Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) at the Indicated Time Points
Description: Hematology parameters were assessed at Entry visit of the extension study, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, and end of study. Change from study AMB115811 Baseline in hemoglobin and MCHC is summarized. AMB115811 Baseline is the last value recorded on or prior to start of study treatment in that study. Change from AMB115811 Baseline was calculated as the value at the indicated visit minus the Baseline value. Participant's final visit in Study AMB115811 was used as the entry visit of this open-label extension study. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). NA indicates that data were not available.
Time Frame: as for outcome 2
Population: Safety (Extension) Population
Measure: Median (Inter-Quartile Range); unit: Grams per Liter (g/L)
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 10
Grams per Liter (g/L)
  Hemoglobin, Entry visit, n=9, 10 | -5.0 [-10 to 2] | -5.5 [-9 to -3]
  Hemoglobin, Month 1, n=7, 10 | -3.0 [-7 to 1] | -6.5 [-9 to -4]
  Hemoglobin, Month 3, n=7, 8 | -7.0 [-25.0 to 8.0] | -10.5 [-14.5 to -1.0]
  Hemoglobin, Month 6, n=5, 6 | -10.0 [-18.0 to 0.0] | -6.5 [-12.0 to -3.0]
  Hemoglobin, Month 9, n=2, 5 | -25.0 [-31.0 to -19.0] | -6.0 [-6.0 to -4.0]
  Hemoglobin, Month 12, n=1, 3 | 21.0 [21.0 to 21.0] | -6.0 [-9.0 to -2.0]
  Hemoglobin, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -11.0 [-11.0 to -11.0]
  Hemoglobin, End of study, n=8, 9 | -10.0 [-15.5 to -2.0] | -8.0 [-11.0 to -2.0]
  MCHC, Entry visit, n=9, 10 | 6.0 [-1.0 to 9.0] | 4.0 [-4.0 to 9.0]
  MCHC, Month 1, n=7, 10 | 5 [-9 to 10] | 1 [-4 to 6]
  MCHC, Month 3, n=7, 8 | 1 [-2 to 4] | 4.5 [-2.5 to 6]
  MCHC, Month 6, n=5, 6 | 3 [1 to 5] | -1.5 [-2 to 0]
  MCHC, Month 9, n=2, 5 | 0.5 [-2 to 3] | -1 [-8 to 0]
  MCHC, Month 12, n=1, 3 | 6.0 [6.0 to 6.0] | -4 [-9 to 5]
  MCHC, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 1 [1 to 1]
  MCHC, End of study, n=8, 9 | -2.0 [-6.0 to 2.5] | -6.0 [-9.0 to -1.0]

4. Primary Outcome: Change From Study AMB115811 Baseline in Hematocrit at the Indicated Time Points
Description: Hematology parameters were assessed at Entry visit of the extension study, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, and end of study. Change from study AMB115811 Baseline in hematocrit is summarized. AMB115811 Baseline is the last value recorded on or prior to start of study treatment in that study. Change from AMB115811 Baseline was calculated as the value at the indicated visit minus the Baseline value. Participant's final visit in study AMB115811 was used as the entry visit of this open-label extension study. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). NA indicates that data were not available.
Time Frame: as for outcome 2
Population: Safety (Extension) Population
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 10
Ratio
  Hematocrit, Entry visit, n=9, 10 | -0.007 [-0.031 to 0.004] | -0.018 [-0.043 to -0.005]
  Hematocrit, Month 1, n=7, 10 | -0.018 [-0.028 to 0.011] | -0.024 [-0.035 to -0.005]
  Hematocrit, Month 3, n=7, 8 | -0.027 [-0.084 to 0.023] | -0.034 [-0.052 to -0.006]
  Hematocrit, Month 6, n=5, 6 | -0.033 [-0.057 to 0.005] | -0.019 [-0.030 to -0.012]
  Hematocrit, Month 9, n=2, 5 | -0.083 [-0.107 to -0.058] | -0.016 [-0.021 to -0.011]
  Hematocrit, Month 12, n=1, 3 | 0.058 [0.058 to 0.058] | -0.009 [-0.036 to 0.001]
  Hematocrit, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -0.034 [-0.034 to -0.034]
  Hematocrit, End of study, n=8, 9 | -0.033 [-0.049 to 0.004] | -0.015 [-0.024 to -0.001]

5. Primary Outcome: Change From Study AMB115811 Baseline in Mean Corpuscle Volume at the Indicated Time Points
Description: Hematology parameters were assessed at Entry visit of the extension study, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, and end of study. Change from study AMB115811 Baseline in mean corpuscle volume is summarized. AMB115811 Baseline is the last value recorded on or prior to start of study treatment in that study. Change from AMB115811 Baseline was calculated as the value at the indicated visit minus the Baseline value. Participant's final visit in study AMB115811 was used as the entry visit of this open-label extension study. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). NA indicates that data were not available.
Time Frame: as for outcome 2
Population: Safety (Extension) Population
Measure: Median (Inter-Quartile Range); unit: Femtoliter (fL)
Groups:
- Ambrisentan 5 mg: Participants received ambrisentan 5 mg tablet OD for 16 weeks in study AMB115811. Upon enrollment in the extension study AMB116457, participants continued to receive ambrisentan 5 mg OD. The dose could be up-titrated to ambrisentan 10 mg OD or adjusted back to ambrisentan 5 mg OD.
Arm/Group | Previous Placebo | Ambrisentan 5 mg
Number analyzed (Participants) | 9 | 10
Femtoliter (fL)
  Mean corpuscle volume, Entry visit, n=9, 10 | -2.0 [-4.0 to -1.0] | -0.5 [-2.0 to 0.0]
  Mean corpuscle volume, Month 1, n=7, 10 | -2.0 [-4.0 to 1.0] | -0.5 [-3.0 to 1.0]
  Mean corpuscle volume, Month 3, n=7, 8 | -2.0 [-6.0 to 1.0] | -1.0 [-4.0 to -0.5]
  Mean corpuscle volume, Month 6, n=5, 6 | -3.0 [-3.0 to 0.0] | -0.5 [-2.0 to 0.0]
  Mean corpuscle volume, Month 9, n=2, 5 | -7.0 [-11.0 to -3.0] | 0.0 [0.0 to 1.0]
  Mean corpuscle volume, Month 12, n=1, 3 | -2.0 [-2.0 to -2.0] | 2.0 [-1.0 to 2.0]
  Mean corpuscle volume, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 1.0 [1.0 to 1.0]
  Mean corpuscle volume, End of study, n=8, 9 | -2.5 [-3.5 to 0.5] | 0.0 [0.0 to 2.0]

6. Primary Outcome: Change From Study AMB115811 Baseline in Red Blood Cell Count and Reticulocytes at the Indicated Time Points
Description: Hematology parameters were assessed at Entry visit of the extension study, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, and end of study. Change from study AMB115811 Baseline in red blood cell count and reticulocytes is summarized. AMB115811 Baseline is the last value recorded on or prior to start of study treatment in that study. Change from AMB115811 Baseline was calculated as the value at the indicated visit minus the Baseline value. Participant's final visit in study AMB115811 was used as the entry visit of this open-label extension study. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). NA indicates that data were not available.
Time Frame: as for outcome 2
Population: Safety (Extension) Population
Measure: Median (Inter-Quartile Range); unit: Tera per Liter (TI/L)
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 10
Tera per Liter (TI/L)
  Red blood cell count, Entry visit , n=9, 10 | -0.20 [-0.30 to 0.20] | -0.15 [-0.40 to -0.10]
  Red blood cell count, Month 1, n=7, 10 | 0.00 [-0.50 to 0.20] | -0.25 [-0.30 to -0.10]
  Red blood cell count, Month 3, n=7, 8 | 0.00 [-0.70 to 0.40] | -0.25 [-0.45 to -0.05]
  Red blood cell count, Month 6, n=5, 6 | -0.30 [-0.70 to 0.10] | -0.15 [-0.30 to 0.00]
  Red blood cell count, Month 9, n=2, 5 | -0.55 [-0.60 to -0.50] | -0.20 [-0.20 to -0.10]
  Red blood cell count, Month 12, n=1, 3 | 0.70 [0.70 to 0.70] | -0.20 [-0.30 to -0.10]
  Red blood cell count, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -0.40 [-0.40 to -0.40]
  Red blood cell count, End of study, n=8, 9 | -0.15 [-0.40 to 0.00] | -0.20 [-0.40 to 0.10]
  Reticulocytes, Entry visit, n=9, 10 | 0.001 [-0.004 to 0.012] | 0.000 [-0.026 to 0.004]
  Reticulocytes, Month 1, n=7, 10 | -0.007 [-0.016 to 0.024] | -0.001 [-0.020 to 0.011]
  Reticulocytes, Month 3, n=7, 8 | 0.001 [-0.016 to 0.011] | -0.001 [-0.022 to 0.011]
  Reticulocytes, Month 6, n=5, 6 | 0.005 [-0.023 to 0.018] | -0.019 [-0.032 to -0.005]
  Reticulocytes, Month 9, n=2, 5 | -0.013 [-0.019 to -0.006] | 0.005 [-0.040 to 0.014]
  Reticulocytes, Month 12, n=1, 3 | -0.032 [-0.032 to -0.032] | 0.017 [-0.003 to 0.027]
  Reticulocytes, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -0.011 [-0.011 to -0.011]
  Reticulocytes, End of study, n=8, 9 | -0.007 [-0.022 to 0.018] | -0.002 [-0.049 to 0.001]

7. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of Potential Clinical Concern at Any Time Post Entry Visit
Description: Blood samples were collected post Entry visit of the extension study and up to end of study for evaluation of the clinical chemistry parameters of alanine amino transferase (ALT), aspartate amino transferase (AST), gamma glutamyl transferase (GGT), and total bilirubin. The clinical chemistry parameters of potential clinical concern high were defined as follows: ALT, AST, GGT >=3 times upper limit of normal (ULN); total bilirubin >=2 times ULN. Participants with both normal and high values were counted once under their worst case (high). Participant's final visit in study AMB115811 was used as the entry visit of this open-label extension study.
Time Frame: Post entry visit of the extension study and up to End of Study (assessed up to approximately 16 months)
Population: Safety (Extension) Population
Measure: Number; unit: Participants
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 10
Participants
  ALT, >clinical concern high | 0 | 0
  AST, >clinical concern high | 0 | 0
  GGT, >clinical concern high | 1 | 0
  Total bilirubin, >clinical concern high | 0 | 0

8. Primary Outcome: Number of Participants With Creatinine Values of Potential Clinical Concern at Any Time Post Entry Visit
Description: Blood samples were collected at Entry visit of the extension study, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, and end of study plus any unscheduled lab tests for creatinine. A creatinine value of potential clinical concern high was defined as >=176.8 micromoles per Liter. Participants with both normal and high values were counted once under their worst case (high). Participant's final visit in study AMB115811 was used as the entry visit of this open-label extension study.
Time Frame: Entry visit of the extension study; Months 1, 3, 6, 9, 12, 15; and End of Study plus any unscheduled lab tests (assessed up to approximately 16 months)
Population: Safety (Extension) Population
Measure: Number; unit: Participants
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 10
Participants | 1 | 0

9. Primary Outcome: Change From Study AMB115811 Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Assessed at the Indicated Time Points
Description: Vital signs including SBP and DBP were assessed at Entry visit of the extension study, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, and end of study. Change from study AMB115811 Baseline in SBP and DBP is summarized. AMB115811 Baseline is the last value recorded on or prior to start of study treatment in that study. Change from AMB115811 Baseline was calculated as the value at the indicated visit minus the Baseline value. Participant's final visit in study AMB115811 was used as the entry visit of this open-label extension study. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). NA indicates that data were not available.
Time Frame: as for outcome 2
Population: Safety (Extension) Population
Measure: Median (Inter-Quartile Range); unit: millimeter of mercury (mmHg)
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 10
millimeter of mercury (mmHg)
  Systolic blood pressure, Entry visit, n=9, 10 | -6.0 [-11.0 to 3.0] | -3.0 [-8.0 to 11.0]
  Systolic blood pressure, Month 1, n=8, 10 | -0.5 [-21.0 to 4.5] | -5.5 [-7.0 to 3.0]
  Systolic blood pressure, Month 3, n=8, 8 | -4.0 [-13.5 to 14.5] | -4.0 [-8.0 to 0.0]
  Systolic blood pressure, Month 6, n=5, 6 | -10.0 [-30.0 to -9.0] | -5.0 [-14.0 to 0.0]
  Systolic blood pressure, Month 9, n=3, 5 | -1.0 [-14.0 to 14.0] | -2.0 [-6.0 to 4.0]
  Systolic blood pressure, Month 12, n=1, 4 | 15.0 [15.0 to 15.0] | -8.5 [-15.5 to 6.5]
  Systolic blood pressure, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -2.0 [-2.0 to -2.0]
  Systolic blood pressure, End of study, n=8, 10 | 2.5 [-14.0 to 12.5] | 1.0 [-5.0 to 5.0]
  Diastolic blood pressure, Entry visit, n=9, 10 | -5.0 [-11.0 to 5.0] | -9.0 [-12.0 to 4.0]
  Diastolic blood pressure, Month 1, n=8, 10 | -9.0 [-17.5 to -3.0] | -7.0 [-10.0 to 4.0]
  Diastolic blood pressure, Month 3, n=8, 8 | -1.0 [-10.5 to 10.0] | -11.0 [-15.5 to -4.0]
  Diastolic blood pressure, Month 6, n=5, 6 | -13.0 [-18.0 to -10.0] | -11.0 [-12.0 to -7.0]
  Diastolic blood pressure, Month 9, n=3, 5 | -5.0 [-7.0 to -4.0] | -7.0 [-12.0 to -5.0]
  Diastolic blood pressure, Month 12, n=1, 4 | 0.0 [0.0 to 0.0] | -9.0 [-16.0 to -5.5]
  Diastolic blood pressure, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -4.0 [-4.0 to -4.0]
  Diastolic blood pressure, End of study, n=8, 10 | -4.0 [-12.0 to 12.0] | -9.5 [-18.0 to -2.0]

10. Primary Outcome: Change From Study AMB115811 Baseline in Heart Rate at the Indicated Time Points
Description: Vital signs including heart rate were assessed at Entry visit of the extension study, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, and end of study. Change from study AMB115811 Baseline in heart rate is summarized. AMB115811 Baseline is the last value recorded on or prior to start of study treatment in that study. Change from AMB115811 Baseline was calculated as the value at the indicated visit minus the Baseline value. Participant's final visit in study AMB115811 was used as the entry visit of this open-label extension study. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). NA indicates that data were not available
Time Frame: as for outcome 2
Population: Safety (Extension) Population
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 10
beats per minute
  Heart rate, Entry visit, n=9, 10 | -2.0 [-17.0 to 5.0] | -7.0 [-17.0 to 1.0]
  Heart rate, Month 1, n=8, 10 | -12.0 [-19.5 to 4.0] | -2.0 [-7.0 to 3.0]
  Heart rate, Month 3, n=8, 8 | -8.5 [-19.0 to 1.5] | -1.0 [-11.0 to 4.5]
  Heart rate, Month 6, n=5, 6 | -19.0 [-24.0 to -14.0] | -3.5 [-6.0 to -1.0]
  Heart rate, Month 9, n=3, 5 | -12.0 [-12.0 to -11.0] | -6.0 [-7.0 to -2.0]
  Heart rate, Month 12, n=1, 4 | -12.0 [-12.0 to -12.0] | -12.5 [-16.5 to -4.5]
  Heart rate, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -11.0 [-11.0 to -11.0]
  Heart rate, End of study, n=8, 10 | -10.5 [-15.0 to 1.0] | 0.5 [-5.0 to 4.0]

11. Primary Outcome: Change From Study AMB115811 Baseline in Weight at the Indicated Time Points
Description: Weight was measured at Entry visit of the extension study, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, and at end of study. Change from study AMB115811 Baseline in weight is summarized. AMB115811 Baseline is the last value recorded on or prior to start of study treatment in that study. Change from AMB115811 Baseline was calculated as the value at the indicated visit minus the Baseline value. Participant's final visit in study AMB115811 was used as the entry visit of this open-label extension study. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). NA indicates that data were not available.
Time Frame: as for outcome 2
Population: Safety (Extension) Population
Measure: Median (Inter-Quartile Range); unit: kilogram (kg)
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 10
kilogram (kg)
  Weight, Entry visit, n=9, 10 | -1.00 [-1.50 to 1.40] | -1.00 [-2.80 to 0.50]
  Weight, Month 1, n=8, 10 | 0.00 [-1.50 to 0.60] | -0.50 [-2.20 to 0.50]
  Weight, Month 3, n=8, 8 | -0.50 [-2.00 to 0.55] | -2.00 [-4.45 to 0.50]
  Weight, Month 6, n=5, 6 | 0.00 [-10.00 to 1.10] | -3.10 [-5.00 to -0.50]
  Weight, Month 9, n=3, 5 | 0.00 [-19.70 to 1.60] | -3.50 [-5.50 to 1.00]
  Weight, Month 12, n=1, 4 | 0.00 [0.00 to 0.00] | -1.15 [-3.25 to 1.00]
  Weight, Month 15, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | -2.50 [-2.50 to -2.50]
  Weight, End of study, n=8, 10 | 0.00 [-1.00 to 0.85] | -0.05 [-2.00 to 1.80]

12. Primary Outcome: Time to First Change in Dose of Open-label Ambrisentan Due to Tolerability Issues in Any Participant
Description: The time to change in dose of ambrisentan or other targeted PAH (pulmonary arterial hypertension) therapeutic agents (prostanoids, PDE-5 inhibitors) due to tolerability issues (e.g. adverse events). Dosing data were collected, but after the study was terminated, not all endpoints listed in the protocol were analyzed, including time to first change in dose of open-label ambrisentan. This decision was documented in the reporting and analysis plan prior to database lock.
Time Frame: From the Entry visit of the extension study up to approximately 16 months
Population: Safety (Extension) Population
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Study AMB115811 Baseline in the 6 Minutes Walking Distance (6MWD) at the Indicated Time Points
Description: The 6-minute walk test was conducted according to the American Thoracic Society guidelines in accordance with local standard operating procedures. 6MWD was measured by a 6-minute walk test. This test measures the distance that a par. can walk in a period of 6 minutes. AMB115811 Baseline was the Week 0 value in that study. Change from study AMB115811 Baseline was calculated as the value at the indicated visit minus the Baseline value. Par.'s final visit in study AMB115811 was used as the entry visit of this extension study. For the Extension study, the visit schedule (Months 1, 3, 6, 9, 12 and 15) was mapped to the visit schedule (Months 5, 7, 10, 13, 16 and 19) for continuity with study AMB115811. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Intent-to-treat (ITT) Population: all par. who were randomized and took at least one dose of study medication in the double-blind phase (placebo or ambrisentan).
Time Frame: During Study AMB115811: Months 0 (Baseline), 1, 2, 3, 4, Early Withdrawal (EW); During Extension Study: Months 1, 3, 6, 9, 12, 15 and at End of Study (assessed up to approximately 20 months)
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: Meters
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 16 | 17
Meters
  (AMB115811) Month 1, n=15, 17 | 5.00 [-1.50 to 16.50] | 14.00 [1.00 to 42.50]
  Month 2, n=14, 16 | 7.50 [-14.50 to 22.50] | 26.25 [3.25 to 61.25]
  Month 3, n=13, 15 | 5.50 [-23.00 to 39.50] | 20.50 [4.00 to 68.00]
  Month 4, n=13, 15 | -10.00 [-32.50 to 20.00] | 25.00 [12.00 to 49.00]
  EW (AMB115811) visit, n=3, 2 | 7.50 [-46.50 to 43.50] | 41.25 [0.00 to 82.50]
  (Extension study) Month 5, n=7, 9 | 0.00 [-15.50 to 40.00] | 51.50 [19.00 to 80.50]
  Month 7, n=7, 8 | -8.00 [-22.50 to 55.00] | 57.50 [23.50 to 88.75]
  Month 10, n=5, 6 | 55.00 [-10.50 to 65.00] | 52.25 [21.00 to 100.00]
  Month 13, n=2, 4 | 8.50 [-5.50 to 22.50] | 33.25 [19.00 to 46.25]
  Month 16, n=1, 4 | 65.00 [65.00 to 65.00] | 47.25 [23.50 to 61.25]
  Month 19, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 69.00 [69.00 to 69.00]
  End of study, n=7, 8 | 30.00 [4.50 to 43.00] | 29.50 [4.00 to 80.25]

14. Secondary Outcome: Change From Study AMB115811 Baseline (BL) in World Health Organization (WHO) Functional Class (FC) at the Indicated Time Points
Description: WHO FC indicates severity of pulmonary arterial hypertension (PAH) and is an adaptation of the New York Heart Association classification, assessed by the investigator. There are 4 grades for WHO FC based on severity of symptoms (Class I = none, Class IV = most severe). Grades mapped to numeric scale 1-4 (i.e. Class IV = 4). WHO FC system links symptoms with activity limitations, allowing clinicians to predict disease progression and prognosis. AMB115811 BL is the last value recorded on or prior to start of study treatment in that study. Change from AMB115811 BL was calculated as the value at the indicated visit minus the BL value (positive change = worsening). Par.'s final visit in AMB115811 was used as entry visit of this ext study. For Ext study, the visit schedule (M1,3,6,9,12 and 15) was mapped to the visit schedule (M5,7,10,13,16 and 19) for continuity with study AMB115811. Only par. available at the specified TP were analyzed (represented by n=X,X in the category title).
Time Frame: During Study AMB115811: Months (M) 0 (Baseline), 1, 2, 3, 4, Early Withdrawal (EW); During Extension (ext) Study: Months 1, 3, 6, 9, 12, 15 and at End of Study (assessed up to approximately 20 months)
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 16 | 17
Scores on a scale
  (AMB115811) Month 1, n=15, 17 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 2, n=14, 16 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 3, n=13, 15 | 0.0 [0.0 to 0.0] | 0.0 [-1.0 to 0.0]
  Month 4, n=13, 15 | 0.0 [0.0 to 0.0] | 0.0 [-1.0 to 0.0]
  EW (AMB115811) visit, n=3, 2 | 0.0 [-1.0 to 0.0] | 0.0 [0.0 to 0.0]
  (Extension study) Month 5, n=8, 10 | 0.0 [0.0 to 0.0] | 0.0 [-1.0 to 0.0]
  Month 7, n=8, 8 | 0.0 [0.0 to 0.5] | 0.0 [-1.0 to 0.0]
  Month 10, n=5, 6 | 0.0 [0.0 to 0.0] | -0.5 [-1.0 to 0.0]
  Month 13, n=3, 5 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 16, n=1, 4 | 0.0 [0.0 to 0.0] | 0.0 [-0.5 to 0.0]
  Month 19, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 0.0 [0.0 to 0.0]
  End of study, n=8, 10 | 0.0 [-0.5 to 0.0] | 0.0 [-1.0 to 0.0]

15. Secondary Outcome: Change From Study AMB115811 Baseline in Borg CR10 Scale (BCR10S) Immediately Following Exercise at the Indicated Time Points
Description: BCR10S score, a rating of perceived exertion, was collected immediately following completion of the 6-minute walk test. Scores range from 0 to 10 (0=nothing at all, 10=extremely strong). If par.'s perception or feeling was stronger than "10", that is "extremely strong", "Maximal" -a larger number could be used, for example 12 or still higher, that is "Absolute maximum"). AMB115811 BL data was calculated as average of 2 BCR10S values obtained following the 2 6MWD tests used in determining the BL 6MWD in that study. If only 1 measurement was available, it was used. Change from AMB115811 BL was calculated as the value at the indicated visit minus the BL value. Par.'s final visit in AMB115811 was used as the entry visit of ext study. For the Ext study, the visit schedule (M1,3,6,9,12 and 15) mapped to the visit schedule (M5,7,10,13,16 and 19) for continuity with AMB115811. Only those par. available at the specified time points were analyzed (represented by n=X,X in the category titles).
Time Frame: as for outcome 14
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 16 | 17
Scores on a scale
  (AMB115811) Month 1, n=15, 17 | 0.00 [-1.00 to 0.75] | -0.40 [-0.50 to 0.00]
  Month 2, n=14, 16 | 0.25 [-0.50 to 1.00] | -0.20 [-1.13 to 1.00]
  Month 3, n=13, 15 | 0.00 [-0.50 to 2.25] | -0.40 [-1.00 to 1.00]
  Month 4, n=13, 15 | 1.00 [-0.50 to 2.50] | -0.50 [-1.50 to 1.00]
  EW (AMB115811) visit, n=3, 2 | 2.00 [-1.50 to 4.00] | -0.25 [-0.50 to 0.00]
  (Extension study) Month 5, n=7, 9 | 0.00 [-0.50 to 1.50] | 1.50 [-0.50 to 2.00]
  Month 7, n=7, 8 | 0.50 [-0.50 to 2.50] | 0.00 [-1.38 to 1.75]
  Month 10, n=5, 6 | 0.50 [0.50 to 1.50] | 0.50 [-1.50 to 1.00]
  Month 13, n=2, 4 | 0.50 [0.50 to 0.50] | 1.00 [-0.75 to 2.75]
  Month 16, n=1, 4 | 0.50 [0.50 to 0.50] | 0.50 [-0.75 to 1.75]
  Month 19, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 1.00 [1.00 to 1.00]
  End of study, n=7, 8 | 1.25 [0.00 to 1.50] | 0.88 [-0.25 to 1.50]

16. Secondary Outcome: Number of Participants With Clinical Worsening of Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Description: Time to clinical worsening of CTEPH was defined as the time from randomization in study AMB115811 to the first occurrence of any of the following events: death (all cause), lung transplantation, hospitalization for CTEPH deterioration, atrial septostomy, addition of parenteral prostanoids, appearance of two or more CTEPH worsening events. Worsening events included: >=20% of decrease in 6MWD; >=1 increase of WHO Functional Classes; worsening right ventricular failure; rapidly progressing cardiogenic, hepatic, or renal failure; refractory systolic hypotension (SBP <85 mmHg).
Time Frame: From randomization up to End of Study for the extension study (assessed up to approximately 20 months)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 16 | 17
Participants | 2 | 0

17. Secondary Outcome: Change From Study AMB115811 Baseline in Quality of Life as Measured by Short Form 36 Health Survey (SF-36)
Description: The SF-36 version 2 is a self-administered, health-related quality of life (QoL) metric. It is a 36-item questionnaire designed to measure 8 domains of functional health status and well-being: physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health as well as 2 summary measures (Physical Health and Mental Health). Each domain is scored from 0 (poorer health) to 100 (better health). Baseline of study AMB115811 was to be used. Change from study AMB115811 Baseline was to be calculated as the value at the indicated visit minus the Baseline value. The SF-36 data were collected, but after the study was terminated, not all endpoints listed in the protocol were analyzed, including the SF-36. This decision was documented in the reporting and analysis plan prior to database lock.
Time Frame: Baseline from study AMB115811 up to End of Study for the extension study (assessed up to approximately 20 months)
Population: ITT Population
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Percent Change From Study AMB115811 Baseline in Plasma N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP)
Description: The ratio to Baseline in NT-proBNP was calculated as the ratio of the value at the specified time-point to the AMB115811 Baseline value and was expressed as a percent change from AMB115811 Baseline. This was done by taking the mean change on the log scale, exponentiating, subtracting 1 and multiplying by 100. Standard deviation (SD) of the logged values (log[SD]) have been presented. AMB115811 Baseline is the last value recorded on or prior to start of study treatment in that study. Participant's final visit in study AMB115811 was used as the entry visit of this open-label extension study. For the Extension study, the visit schedule (Months 1, 3, 6, 9, 12 and 15) was mapped to the visit schedule (Months 5, 7, 10, 13, 16 and 19) for continuity with study AMB115811. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). NA indicates that data were not available.
Time Frame: as for outcome 13
Population: ITT Population
Measure: Geometric Mean (Standard Deviation); unit: Percent change
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 16 | 17
Percent change
  (AMB115811) Month 1, n=13, 15 | 43.6 (0.41) | -15.8 (0.36)
  Month 2, n=13, 15 | 12.4 (0.49) | -23.3 (0.59)
  Month 3, n=12, 14 | 12.4 (0.59) | -21.9 (0.61)
  Month 4, n=12, 14 | 14.1 (0.55) | -29.4 (0.50)
  EW (AMB115811) visit, n=3, 2 | 35.7 (0.69) | -14.9 (0.31)
  (Extension study) Month 5, n=8, 10 | -34.7 (1.22) | -24.5 (0.69)
  Month 7, n=8, 8 | 3.3 (0.64) | -32.5 (0.73)
  Month 10, n=5, 6 | -36.5 (0.86) | -20.1 (0.78)
  Month 13, n=3, 5 | -8.6 (0.60) | 7.7 (0.79)
  Month 16, n=1, 4 | -62.4 (NA) — The standard deviation could not be calculated as the number of participants analyzed was 1. | -2.8 (1.15)
  Month 19, n=0, 1 | NA (NA) — No participants were analyzed at this time point. | 43.1 (NA) — The standard deviation could not be calculated as the number of participants analyzed was 1
  End of study, n=8, 9 | -13.2 (0.72) | -41.7 (0.86)

19. Secondary Outcome: Change From Start of Ambrisentan Treatment in 6 Minutes Walking Distance at the Indicated Time Points
Description: The 6 minute walk distance data in a previous outcome measure were also analyzed as change from start of ambrisentan treatment. As participants started to receive ambrisentan treatment in two studies, two different time points for start of ambrisentan treatment were used for this analysis. For participants who received ambrisentan treatment in Study AMB115811, the Baseline for that study was used. For participants who received placebo in Study AMB115811, entry visit of the Extension study was defined as Baseline. Change from start of ambrisentan was calculated as the value at the indicated visit minus the start of ambrisentan value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category title).
Time Frame: Previous Placebo: Months 0 (Entry visit of the extension), 1, 3, 6, 9, 12; Previous Ambrisentan: Month 0 (Baseline of study AMB115811), 1, 2, 3, 4, Early Withdrawal (EW) (AMB115811), 5, 7, 10, 13, 16, 19; and at End of Study
Population: ITT Population. Placebo arm: includes par. who received ambrisentan treatment during extension study
Measure: Median (Inter-Quartile Range); unit: Meters
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 17
Meters
  Month 1, n=7, 17 | 20.00 [15.00 to 30.00] | 14.00 [1.00 to 42.50]
  Month 2, n=0, 16 | NA [NA to NA] — No participants were analyzed at this time point. | 26.25 [3.25 to 61.25]
  Month 3, n=7, 15 | 20.00 [15.00 to 35.00] | 20.50 [4.00 to 68.00]
  Month 4, n= 0, 15 | NA [NA to NA] — No participants were analyzed at this time point. | 25.00 [12.00 to 49.00]
  EW (AMB115811), n=0, 2 | NA [NA to NA] — No participants were analyzed at this time point. | 41.25 [0.00 to 82.50]
  Month 5, n=0, 9 | NA [NA to NA] — No participants were analyzed at this time point. | 51.50 [19.00 to 80.50]
  Month 6, n=5, 0 | 45.00 [27.00 to 60.00] | NA [NA to NA] — No participants were analyzed at this time point.
  Month 7, n=0, 8 | NA [NA to NA] — No participants were analyzed at this time point. | 57.50 [23.50 to 88.75]
  Month 9, n=2, 0 | 32.50 [5.00 to 60.00] | NA [NA to NA] — No participants were analyzed at this time point.
  Month 10, n=0, 6 | NA [NA to NA] — No participants were analyzed at this time point. | 52.25 [21.00 to 100.00]
  Month 12, n=1, 0 | 45.00 [45.00 to 45.00] | NA [NA to NA] — No participants were analyzed at this time point.
  Month 13, n=0, 4 | NA [NA to NA] — No participants were analyzed at this time point. | 33.25 [19.00 to 46.25]
  Month 16, n=0, 4 | NA [NA to NA] — No participants were analyzed at this time point. | 47.25 [23.50 to 61.25]
  Month 19, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 69.00 [69.00 to 69.00]
  End of study, n=7, 8 | 37.00 [0.00 to 60.00] | 29.50 [4.00 to 80.25]

20. Secondary Outcome: Change From Start of Ambrisentan Treatment in World Health Organization (WHO) Functional Class (FC) at the Indicated Time Points
Description: The WHO functional class data in a previous outcome measure were also analyzed as change from start of ambrisentan treatment. There are 4 grades for WHO FC based on severity of symptoms of pulmonary arterial hypertension (Class I = none, Class IV = most severe). Grades mapped to numeric scale 1-4 (i.e. Class IV = 4). As participants started to receive ambrisentan treatment in two studies, two different time points for start of ambrisentan treatment were used for this analysis. For participants who received ambrisentan treatment in Study AMB115811, the Baseline for that study was used. For participants who received placebo in Study AMB115811, entry visit of the Extension study was defined as Baseline. Change from start of ambrisentan was calculated as the value at the indicated visit minus the start of ambrisentan value (positive change = worsening). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: as for outcome 19
Population: ITT Population. Placebo arm: includes par. who received ambrisentan treatment during extension study
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 17
Scores on a scale
  Month 1, n=8, 17 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Month 2, n=0, 16 | NA [NA to NA] — No participants were analyzed at this time point. | 0.0 [0.0 to 0.0]
  Month 3, n=8, 15 | 0.0 [0.0 to 0.0] | 0.0 [-1.0 to 0.0]
  Month 4, n= 0, 15 | NA [NA to NA] — No participants were analyzed at this time point. | 0.0 [-1.0 to 0.0]
  EW (AMB115811), n=0, 2 | NA [NA to NA] — No participants were analyzed at this time point. | 0.0 [0.0 to 0.0]
  Month 5, n=0, 10 | NA [NA to NA] — No participants were analyzed at this time point. | 0.0 [-1.0 to 0.0]
  Month 6, n=5, 0 | 0.0 [0.0 to 0.0] | NA [NA to NA] — No participants were analyzed at this time point.
  Month 7, n=0, 8 | NA [NA to NA] — No participants were analyzed at this time point. | 0.0 [-1.0 to 0.0]
  Month 9, n=3, 0 | 0.0 [0.0 to 0.0] | NA [NA to NA] — No participants were analyzed at this time point.
  Month 10, n=0, 6 | NA [NA to NA] — No participants were analyzed at this time point. | -0.5 [-1.0 to 0.0]
  Month 12, n=1, 0 | 0.0 [0.0 to 0.0] | NA [NA to NA] — No participants were analyzed at this time point.
  Month 13, n=0, 5 | NA [NA to NA] — No participants were analyzed at this time point. | 0.0 [0.0 to 0.0]
  Month 16, n=0, 4 | NA [NA to NA] — No participants were analyzed at this time point. | 0.0 [-0.5 to 0.0]
  Month 19, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 0.0 [0.0 to 0.0]
  End of study, n=8, 10 | 0.0 [0.0 to 0.0] | 0.0 [-1.0 to 0.0]

21. Secondary Outcome: Change From Start of Ambrisentan Treatment in Borg CR10 Scale (BCR10S) Immediately Following Exercise at the Indicated Time Points
Description: The BCR10S data in a previous outcome measure were also analyzed as change from start of ambrisentan treatment. BCR10S score, a rating of perceived exertion, ranges from 0 to 10 (0=nothing at all, 10 extremely strong). If par.'s perception or feeling was stronger than "10", a larger number could be used. As participants started to receive ambrisentan treatment in two studies, two different time points for start of ambrisentan treatment were used for this analysis. For participants who received ambrisentan treatment in Study AMB115811, the Baseline for that study was used. For participants who received placebo in Study AMB115811, entry visit of the Extension study was defined as Baseline. Change from start of ambrisentan was calculated as the value at the indicated visit minus the start of ambrisentan value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category title).
Time Frame: as for outcome 19
Population: ITT Population. Placebo arm: includes par. who received ambrisentan treatment during extension study
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 17
Scores on a scale
  Month 1, n=7, 17 | 0.00 [-1.00 to 1.00] | -0.40 [-0.50 to 0.00]
  Month 2, n=0, 16 | NA [NA to NA] — No participants were analyzed at this time point. | -0.20 [-1.13 to 1.00]
  Month 3, n=7, 15 | 0.00 [0.00 to 1.00] | -0.40 [-1.00 to 1.00]
  Month 4, n= 0, 15 | NA [NA to NA] — No participants were analyzed at this time point. | -0.50 [-1.50 to 1.00]
  EW (AMB115811), n=0, 2 | NA [NA to NA] — No participants were analyzed at this time point. | -0.25 [-0.50 to 0.00]
  Month 5, n=0, 9 | NA [NA to NA] — No participants were analyzed at this time point. | 1.50 [-0.50 to 2.00]
  Month 6, n=5, 0 | 1.00 [1.00 to 2.00] | NA [NA to NA] — No participants were analyzed at this time point.
  Month 7, n=0, 8 | NA [NA to NA] — No participants were analyzed at this time point. | 0.00 [-1.38 to 1.75]
  Month 9, n=2, 0 | 0.50 [-1.00 to 2.00] | NA [NA to NA] — No participants were analyzed at this time point.
  Month 10, n=0, 6 | NA [NA to NA] — No participants were analyzed at this time point. | 0.50 [-1.50 to 1.00]
  Month 12, n=1,0 | 1.00 [1.00 to 1.00] | NA [NA to NA] — No participants were analyzed at this time point.
  Month 13, n=0, 4 | NA [NA to NA] — No participants were analyzed at this time point. | 1.00 [-0.75 to 2.75]
  Month 16, n=0, 4 | NA [NA to NA] — No participants were analyzed at this time point. | 0.50 [-0.75 to 1.75]
  Month 19, n=0, 1 | NA [NA to NA] — No participants were analyzed at this time point. | 1.00 [1.00 to 1.00]
  End of study, n=7, 8 | 0.00 [-1.00 to 1.00] | 0.88 [-0.25 to 1.50]

22. Secondary Outcome: Percent Change From Start of Ambrisentan Treatment in Plasma N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP)
Description: The NT-proBNP data in a previous outcome measure were also analyzed as change from start of ambrisentan treatment. The ratio to start of ambrisentan in NT-proBNP was calculated as the ratio of the value at the specified time-point to the start of ambrisentan value and was expressed as a percent change from start of ambrisentan. This was done by taking the mean change on the log scale, exponentiating, subtracting 1 and multiplying by 100. Standard deviation (SD) of the logged values (log[SD]) have been presented. As par. started to receive ambrisentan treatment in 2 studies, 2 different time points for start of ambrisentan treatment were used for this analysis. For par. who received ambrisentan treatment in study AMB115811, the Baseline for that study was used. For par. who received placebo in Study AMB115811, entry visit of the Extension study was defined as Baseline. Only those par. available at the specified time points were analyzed (represented by n=X, X in the category title).
Time Frame: as for outcome 19
Population: ITT Population. Placebo arm: includes par. who received ambrisentan treatment during extension study
Measure: Geometric Mean (Standard Deviation); unit: Percent change
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 9 | 17
Percent change
  Month 1, n=8, 15 | -49.5 (1.40) | -15.8 (0.36)
  Month 2, n=0, 15 | NA (NA) — No participants were analyzed at this time point. | -23.3 (0.59)
  Month 3, n=8, 14 | -20.1 (0.86) | -21.9 (0.61)
  Month 4, n= 0, 14 | NA (NA) — No participants were analyzed at this time point. | -29.4 (0.50)
  EW (AMB115811), n=0, 2 | NA (NA) — No participants were analyzed at this time point. | -14.9 (0.31)
  Month 5, n=1, 10 | NA (NA) — Month 5 for the Previous Placebo arm was an unscheduled lab assessment; therefore, the value was entered as NA for the 1 participant at this time point. | -24.5 (0.69)
  Month 6, n=5, 0 | -53.5 (1.22) | NA (NA) — No participants were analyzed at this time point.
  Month 7, n=0, 8 | NA (NA) — No participants were analyzed at this time point. | -32.5 (0.73)
  Month 9, n=3, 1 | -11.2 (0.71) | NA (NA) — Month 9 for the Previous ambrisentan arm was an unscheduled lab assessment; therefore, the value was entered as NA for the 1 participant at this time point.
  Month 10, n=0, 6 | NA (NA) — No participants were analyzed at this time point. | -20.1 (0.78)
  Month 12, n=1, 0 | -67.9 (NA) — The standard deviation could not be calculated as the number of participants analyzed was 1. | NA (NA) — No participants were analyzed at this time point.
  Month 13, n=0, 5 | NA (NA) — No participants were analyzed at this time point. | 7.7 (0.79)
  Month 16, n=0, 4 | NA (NA) — No participants were analyzed at this time point. | -2.8 (1.15)
  Month 19, n=0, 1 | NA (NA) — No participants were analyzed at this time point. | 43.1 (NA) — The standard deviation could not be calculated as the number of participants analyzed was 1.
  End of study, n=8, 9 | -30.5 (0.85) | -41.7 (0.86)

23. Secondary Outcome: Time to First Change in Dose of Open-label Ambrisentan Due to Deterioration of Clinical Conditions in Any Participant
Description: The time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to deterioration of clinical condition. Dosing data were collected, but after the study was terminated, not all endpoints listed in the protocol were analyzed, including time to first change in dose of open-label ambrisentan. This decision was documented in the reporting and analysis plan prior to database lock.
Time Frame: From Entry visit of the extension study up to End of Study (assessed up to approximately 16 months)
Population: Safety (Extension) Population
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Time to First Addition of Another Targeted PAH Therapeutic Agent Due to Deterioration of Clinical Condition or Lack of Beneficial Effect With Previous Therapy in Any Participant
Description: The time to addition of another targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to the following reasons:
  Deterioration of clinical condition; Lack of beneficial effect with previous therapy (not reaching set treatment goals). PAH therapies were collected, but after the study was terminated, not all endpoints listed in the protocol were analyzed, including time to first addition of another targeted PAH therapeutic agent. This decision was documented in the reporting and analysis plan prior to database lock.
Time Frame: From Entry visit of the extension study up to End of Study (assessed up to approximately 16 months)
Population: Safety (Extension) Population.
Arm/Group | Previous Placebo | Previous Ambrisentan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) will include AEs up to 30 days after their last dose, assessed up to approximately 16 months.
Description: TEAEs are reported for the Safety (Extension) Population. TEAEs are: a) new events that started during the extension study. For par. withdrawn from the study, TEAEs included AEs up to 30 days after last dose b) ongoing AEs that started before the extension study but were either not reported in study AMB115811 or worsened during the extension study.
Arm/Group | Previous Placebo | Previous Ambrisentan
Serious Adverse Events (participants affected / at risk) | 3/9 | 0/10
Other Adverse Events (participants affected / at risk) | 8/9 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Previous Placebo (N=9) | Previous Ambrisentan (N=10)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Implant site extravasation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Previous Placebo (N=9) | Previous Ambrisentan (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hyperthermia (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 0
Bacteriuria (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.